CLINICAL TRIAL: NCT06434987
Title: Impact of Retrograde Inferior Vena Cava Perfusion on Gastrointestinal Function in Patients Undergoing Surgical Repair for Acute Type A Aortic Dissection: A Study Protocol and Prospective Evaluation.
Brief Title: Impact of RIVP on GI Function in Patients Undergoing Surgical Repair for ATAAD
Status: Recruiting | Type: Observational
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-KY-215-01
Record Dates: First submitted 2024-05-15; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-04

CONDITIONS: Type A Aortic Dissection
Keywords: Acute Type A Aortic Dissection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ATAAD patients undergoing Cardiopulmonary Bypass (CPB) with RIVP: ACP+RIVP under mild to moderate hypothermia
  Interventions: Procedure: Retrograde Inferior Vena Cava Perfusion
- ATAAD patients undergoing Cardiopulmonary Bypass (CPB) without RIVP: ACP only under mild to moderate hypothermia.
  Interventions: Procedure: Antegrade cerebral perfusion

INTERVENTIONS:
Procedure: Retrograde Inferior Vena Cava Perfusion — Retrograde inferior vena cava (RIVP) involves perfusing oxygenated blood into the inferior vena cava, which then flows towards the viscera, abdominal organs and lower extremities. By maintaining perfusion to these regions during cardiopulmonary bypass (CPB) and induced hypothermia, Retrograde inferior vena cava (RIVP) helps mitigate the risk of ischemic injury to the abdominal organs. Following the initiation of total cardiopulmonary bypass, the body temperature will be gradually lowered to achieve deep-moderate hypothermia ( 24-38°C). This procedure will involve the combination of selective antegrade cerebral perfusion and retrograde inferior vena cava perfusion. Antegrade perfusion will be maintained at a flow rate of 5-7mL/min/kg, while retrograde perfusion will be regulated to sustain the required pumm pressure and blood flow.
  Groups: ATAAD patients undergoing Cardiopulmonary Bypass (CPB) with RIVP
Procedure: Antegrade cerebral perfusion — After mild to moderate hypothermia is achieved, a cannula will be inserted into the right axillary artery, brachiocephalic or innominate artery to provide continuous flow to the brain. A flow rate of 5-7mL/min/kg will be maintained.
  Groups: ATAAD patients undergoing Cardiopulmonary Bypass (CPB) without RIVP

SUMMARY:
Acute Type A Aortic Dissection (ATAAD) is a serious medical condition that requires immediate surgical intervention. The repair of Acute Type A Aortic Dissection (ATAAD) combines different surgical procedures, including the use of Cardiopulmonary Bypass (CPB). This study focuses on the gastrointestinal (GI) system and the complications arising in the gastrointestinal (GI) system as a result of this procedure. Retrograde Inferior Vena Cava Perfusion (RIVP) is a technique used during Cardiopulmonary Bypass (CPB) that could show potential in mitigating latent gastrointestinal (GI) complications. The study aims to evaluate the effectiveness of Retrograde Inferior Vena Cava Perfusion (RIVP) in patients receiving Acute Type A Aortic Dissection (ATAAD) repair with Cardiopulmonary Bypass (CPB) in reducing Ischemic Reperfusion (IR) injury and inflammatory responses that affect gastrointestinal (GI) integrity. It intends to compare the postoperative gastrointestinal (GI) complications and long-term gastrointestinal (GI) function between patients treated with Antegrade Cerebral Perfusion (ACP) and Retrograde Inferior Vena Cava Perfusion (RIVP), and those treated with Antegrade Cerebral Perfusion (ACP) alone. The patients will be placed in their respective groups as per the decision of the surgeons, perfusionists, and the condition of the patient. Data collection will be facilitated by a comprehensive Case Report Form (CRF). This pilot study, guided by established methodologies, places the study's sample size at 30 to ensure statistical reliability and prevent resource wastage. Through this approach of sample collection, baseline data collection, peri-operative data recording, and follow-up assessments, the study aims to shed light on the impact of Retrograde Inferior Vena Cava Perfusion (RIVP) during Acute Type A Aortic Dissection (ATAAD) repair on gastrointestinal (GI) complications and systemic/intestinal inflammation. The integration of specialized Case Report Forms (CRFs) and structured questionnaires ensures standardized data collection and management, while prioritizing patient confidentiality. The study's data analysis, powered by R software, will provide valuable insights into the efficacy of Retrograde Inferior Vena Cava Perfusion (RIVP) in enhancing clinical outcomes and improving patient's prognosis in the surgical treatment of Acute Type A Aortic Dissection (ATAAD).

DETAILED DESCRIPTION:
Retrograde Inferior Vena Cava Perfusion ( RIVP) is a adjunct technique used in surgery during the repair of Acute Type A Aortic Dissection (ATAAD). This procedure generally involves perfusing oxygenated blood into the inferior vena cava, directing it toward the visceral organs and lower extremities. This technique plays an important role in reducing the risk of ischemic injury to these vital regions during deep hypothermic circulatory arrest (DHCA) when combined with Antegrade Cerebral Perfusion (ACP).

Recent study showed that the use of Retrograde Inferior Vena Cava Perfusion (RIVP), in conjunction with Antegrade Cerebral Perfusion (ACP), may lead to lower rates of organ dysfunction in the lower body, reduced mortality and shorter Cardiopulmonary Bypass (CPB) duration. It has also been associated with maintaining higher higher body temperature during circulatory arrest which may be beneficial for the overall patient well-being.

However, despite these promising results , there is a need for further research to explore the scientific impact of Retrograde Inferior Vena Cava Perfusion (RIVP) on gastrointestinal function during and after Acute Type A Aortic Dissection (ATAAD) repair. Gastrointestinal complications are a crucial aspect of a patients outcomes, and more often neglected. Understanding the relationship between Retrograde Inferior Vena Cava Perfusion (RIVP) and these complications may be essential and have the potential to lead better prognosis among patients, resulting in improved outcomes.

In summary, Retrograde Inferior Vena Cava Perfusion (RIVP) is a valuable technique that helps protect abdominal organs and lower extremities during Acute Type A Aortic Dissection (ATAAD) surgery. While it shows promise in improving patient outcomes, ongoing research is necessary to comprehensively assess its effect on gastrointestinal function, thus optimizing its use in the surgical management of Acute Type A Aortic Dissection (ATAAD).

This study is designed as a single centered, prospective, cohort study with an exploratory framework. The study will be conducted at the Second Affiliated Hospital of Nanjing Medical University Cardiovascular Center. This study will focus on patients undergoing Acute Type A Aortic Dissection (ATAAD) repair with or without Retrograde Inferior Vena Cava Perfusion (RIVP). Patients will be assigned to these groups based on surgical and patient specific criteria in the ratio 1:1 and will follow patients in the Cardiovascular Critical Care Unit ( CCU) pre-operatively. Group A will receive selective ACP+RIVP, while group B will receive ACP alone under mild to moderate hypothermia. As per the general rule of thumb, the study anticipates to recruit up to 30 patients for the pilot study in total. 15 in each group.

Patients will undergo diagnostic assessments to confirm diagnosis of Acute Type A Aortic Dissection (ATAAD) and depending on urgency they will proceed either to surgery or Cardiovascular Critical Care Unit (CCU). Informed consent will be obtained, but this will in no way delay the treatment protocol for the patients. In case of urgent surgery, a surgical fellow will obtain the consent. Patients can withdraw without repercussions and no replacements will be sought.

All data will be collected and recorded systematically in a well drafted case report form. A protocol has been written to conduct this study and we have followed the SPIRITS guidelines. Any changes in the protocol will be timely reported and adjusted.

We will collect blood samples at specific time intervals, pre operatively (PO1), post operatively day 1 (PO2), day 3 (PO3), day 7 (PO4). The study will include biomarker evaluation: CRP, intestinal barrier indicators ( D-amine oxidase(DAO), Fatty Acid Binding Protein 2 (FABP2), D-Lactate, Endotoxins) and 12 cytokine panel.

All baseline data ranging from clinical parameters, anthropometric data, baseline gastrointestinal (GI) assessment and clinical data will be obtained before surgery and recorded in the case report form.

Peri operative data, duration of Cardiopulmonary Bypass (CPB), duration of deep hypothermic circulatory arrest (DHCA), cross clamp time, surgery time, number of units of whole blood, fresh frozen plasma, pooled platelets and cryoprecipitate administered will be collected within the surgical room by the perfusionist and the anesthesiologist.

A prospective longitudinal study will assess long term gastrointestinal (GI) dysfunction post surgery through follow up methods such as outpatient, Wechat application, in hospital or telephone based follow up evaluation at specified intervals (1,3,6,12 months) post hospital discharge. A meticulously drafted questionnaire will be used as a tool for assessment.

To establish presence of gut barrier dysfunction, the investigators will look at the specific patterns or deviation in values of the biomarkers from the normal or baseline levels. An increase in pro-inflammatory cytokines may suggest an inflammatory response associated with gut barrier dysfunction. Elevated levels of D- Lactate, Fatty Acid Binding Protein 2 (FABP2) and endotoxins and decreased activity levels of D-amine oxidase (DAO) could suggest gut barrier dysfunction.

The investigators will perform comprehensive statistical analysis to evaluate continuous variables, like inflammatory markers. This includes calculating the mean, standard deviation and interquartile range for values related to C- reactive protein (CRP), cytokines and intestinal barrier markers. The investigators will use the t-test to analyze differences in these variables. For ordinal data from the Case Report Form (CRF) and follow up questionnaire, wilcoxon rank sun test for hypothesis testing will be used. Categorical data will be presented as percentages , and the differences in these categories will be assessed using the chi-squared test. To handle data at multiple time points, ANOVA will be used to assess variance. When dealing with multiple dependant variables like various cytokine levels simultaneously , the investigators will employ a multivariate analysis of variance. We will consider results statistically significant if the p value is <0.05, in lone with established research and data analysis practices.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing ATAAD repair under CPB.
2. Age: 18-70 years
3. Give consent

Exclusion Criteria:

1. Variables that can influence gut microbiome like antibiotics or probiotics 2 weeks prior to surgery
2. On chemotherapy
3. Evidence of pre-operative malperfusion of the GI system
4. Presence of GI any pathology (IBD,GERD,PU)
5. Continuous enteral feeding prior to surgery
6. Refuse to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study groups with be patients undergoing ATAAD repair under CPB with and without RIVP. This is a cohort study and the patients will not be assigned any specific group randomly or by a computer. The patients will be placed in their respective groups as per the decision of the surgeons, perfusionist and the condition of the patient. Patients admitted through the emergency department will be initially enrolled into the cardiovascular department and subsequently invited to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-12-25 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
RIVP will reduce post operative GI disturbances and gut barrier dysfunction. | Pre operatively, Post -operative day 1 ,day 2, day 3 and day 7
  Patients undergoing CPB with RIVP may have a better prognosis and less incidence of long term GI disturbance as compared to those patients undergoing CPB without RIVP. Measurement tools: 1. Biomarkers; levels of D-Lactate, FABP2 ( Fatty Acid Binding Protein 2), endotoxins and DAO (Diamine Oxidase). Measurement method: Samples of blood will be analyzed using ELISA ( Enzyme Linked Immunosorbent Assay)
Inflammatory response will be possibly reduced in those undergoing RIVP | Pre operatively, Post -operative day 1 ,day 2, day 3 and day 7
  Measurements: C-Reactive protein (CRP) and 12 cytokine panel. Method: blood samples will be analyzed using immunoassays
Gastrointestinal assessment and long term gastrointestinal dysfunction. | Follow up questionaires will be addressed at 1,3,6 and 12 months post hospital discharge. Follow up will be outpatient visits, telephone based calls and interviews, wechat application at the specified intervals
  Measurement tools: clinical assessment for gastrointestinal function and questionnaire. Special formulated case report forms will contain a detailed questionnaire assessing the quality of life and gastrointestinal function. Method: Baseline gastrointestinal function will be assessed pre opratively and follow up questionnaire post operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Qing Guo Li, Study Chair — The Second Hospital of Nanjing Medical University; Sanaa Azim, Principal Investigator — The Second Affiliate Hospital of Nanjing Medical University
Locations (1):
- The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Harris KM, Nienaber CA, Peterson MD, Woznicki EM, Braverman AC, Trimarchi S, Myrmel T, Pyeritz R, Hutchison S, Strauss C, Ehrlich MP, Gleason TG, Korach A, Montgomery DG, Isselbacher EM, Eagle KA. Early Mortality in Type A Acute Aortic Dissection: Insights From the International Registry of Acute Aortic Dissection. JAMA Cardiol. 2022 Oct 1;7(10):1009-1015. doi: 10.1001/jamacardio.2022.2718. PMID 36001309
- [Background] Salomon J, Ericsson A, Price A, Manithody C, Murry DJ, Chhonker YS, Buchanan P, Lindsey ML, Singh AB, Jain AK. Dysbiosis and Intestinal Barrier Dysfunction in Pediatric Congenital Heart Disease Is Exacerbated Following Cardiopulmonary Bypass. JACC Basic Transl Sci. 2021 Mar 3;6(4):311-327. doi: 10.1016/j.jacbts.2020.12.012. eCollection 2021 Apr. PMID 33997519
- [Background] Cheng LK, O'Grady G, Du P, Egbuji JU, Windsor JA, Pullan AJ. Gastrointestinal system. Wiley Interdiscip Rev Syst Biol Med. 2010 Jan-Feb;2(1):65-79. doi: 10.1002/wsbm.19. PMID 20836011
- [Background] Sarkar M, Prabhu V. Basics of cardiopulmonary bypass. Indian J Anaesth. 2017 Sep;61(9):760-767. doi: 10.4103/ija.IJA_379_17. PMID 28970635
- [Background] Halter J, Steinberg J, Fink G, Lutz C, Picone A, Maybury R, Fedors N, DiRocco J, Lee HM, Nieman G. Evidence of systemic cytokine release in patients undergoing cardiopulmonary bypass. J Extra Corpor Technol. 2005 Sep;37(3):272-7. PMID 16350379
- [Background] Typpo KV, Larmonier CB, Deschenes J, Redford D, Kiela PR, Ghishan FK. Clinical characteristics associated with postoperative intestinal epithelial barrier dysfunction in children with congenital heart disease. Pediatr Crit Care Med. 2015 Jan;16(1):37-44. doi: 10.1097/PCC.0000000000000256. PMID 25162512
- [Background] Yan TD, Bannon PG, Bavaria J, Coselli JS, Elefteriades JA, Griepp RB, Hughes GC, LeMaire SA, Kazui T, Kouchoukos NT, Misfeld M, Mohr FW, Oo A, Svensson LG, Tian DH. Consensus on hypothermia in aortic arch surgery. Ann Cardiothorac Surg. 2013 Mar;2(2):163-8. doi: 10.3978/j.issn.2225-319X.2013.03.03. PMID 23977577
- [Background] Safi HJ, Miller CC 3rd, Lee TY, Estrera AL. Repair of ascending and transverse aortic arch. J Thorac Cardiovasc Surg. 2011 Sep;142(3):630-3. doi: 10.1016/j.jtcvs.2010.11.015. Epub 2011 Jan 26. PMID 21269650
- [Background] Ehrlich M, Fang WC, Grabenwoger M, Cartes-Zumelzu F, Wolner E, Havel M. Perioperative risk factors for mortality in patients with acute type A aortic dissection. Circulation. 1998 Nov 10;98(19 Suppl):II294-8. PMID 9852917
- [Background] Ziyaeifard M, Alizadehasl A, Massoumi G. Modified ultrafiltration during cardiopulmonary bypass and postoperative course of pediatric cardiac surgery. Res Cardiovasc Med. 2014 May;3(2):e17830. doi: 10.5812/cardiovascmed.17830. Epub 2014 Apr 1. PMID 25478538
- [Background] Lin J, Qin Z, Liu X, Xiong J, Wu Z, Guo Y, Kang D, Du L. Retrograde inferior vena caval perfusion for total aortic arch replacement surgery: a randomized pilot study. BMC Cardiovasc Disord. 2021 Apr 20;21(1):193. doi: 10.1186/s12872-021-02002-9. PMID 33879045